CLINICAL TRIAL: NCT04751071
Title: The Phosphodiesterase 4 Inhibitor Roflumilast as an Adjunct to Antidepressants in Major Depressive Disorder Patients. Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Phosphodiesterase 4 Inhibitor Roflumilast as an Adjunct to Antidepressants in Major Depressive Disorder Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2021NEUR2
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roflumilast (Active Comparator): Roflumilast 500 µg tablet plus standard therapy
  Interventions: Drug: Roflumilast 500Mcg Tab
- Placebo (Placebo Comparator): placebo tablet plus standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast 500Mcg Tab — Roflumilast 500µg tablet once daily for 6 weeks plus the standard therapy
  Arms: Roflumilast
Drug: Placebo — Placebo tablet once daily for 6 weeks plus the standard therapy
  Arms: Placebo

SUMMARY:
n pre-clinical studies and early-stage clinical trials, PDE4 inhibitors such as rolipram have been shown to enhance memory. They also improve depressive-like behaviors induced by chronic unpredictable mild stress, lipopolysaccharide, or ethanol abstinence . Consequently, it is reasonable to believe that PDE4 is a potential target for treatment of the comorbidity of depression and AD.The aim of the current study is to evaluate the potential adjunct antidepressant effect of the Phosphodiesterase-4 Inhibitor Roflumilast in adult patients with MDD.

DETAILED DESCRIPTION:
Phosphodiesterase-4 (PDE4), an important member of the PDE superfamily, is a key regulator of intracellular cyclic AMP (cAMP) level. As the second messenger, cAMP activates protein kinase A, which phosphorylates the subsequent downstream cAMP-response element binding (CREB) protein. In the central nervous system, this signaling cascade exerts both pre- and post-synaptic effects and is essential for a variety of cellular functions, including neurotransmitter release and neuroprotection. Inhibition of PDE4 prevents cAMP breakdown, which is well recognized as the mechanism by which PDE4 inhibitors can treat impaired memory linked to several brain disorders. In pre-clinical studies and early-stage clinical trials, PDE4 inhibitors such as rolipram have been shown to enhance memory. They also improve depressive-like behaviors induced by chronic unpredictable mild stress, lipopolysaccharide, or ethanol abstinence . Consequently, it is reasonable to believe that PDE4 is a potential target for treatment of the comorbidity of depression and AD.

The aim of the current study is to evaluate the potential adjunct antidepressant effect of Roflumilast in adult patients with MDD. Furthermore, we will assess the relationship between HAM-D score and BDNF as well as their role as a therapeutic targets of MDD.

ELIGIBILITY:
Inclusion Criteria:

• Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 20 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical condition
* Patients with history of seizures
* Patients with history of receiving Electroconvulsive therapy (ECT)
* Patients with inflammatory disorders
* Patients with allergy or contraindications to the used medications
* Patients with finally pregnant or lactating females
* Cardiovascular disorders
* Severe renal impairment: creatinine clearance of ≤ 25 ml/min
* Moderate or severe hepatic impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | 6 weeks
  The principal measure of the outcome was the 17-items Effect on Hamilton Depression rating scale score. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as Effect on Hamilton Depression rating scale total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the Effect on Hamilton Depression rating scale total score.

SECONDARY OUTCOMES:
Effect on biological markers | 6 weeks
  Serum level of brain derived neurotrophic factor (BDNF)
Effect on biological markers | 6 weeks
  Serum level of cAMP response element-binding protein (CREB)
Effect on biological markers | 6 weeks
  Serum level of SEROTONIN
Effect on biological markers | 6 weeks
  Serum level of tumor necrosis factor alpha (TNF-α)
Effect on biological markers | 6 weeks
  Serum level of Interleukin-6 (IL-6)
Effect on biological markers | 6 weeks
  Serum level of Nuclear factor kappa

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibeen Elkom, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF